CLINICAL TRIAL: NCT04936269
Title: Psychometric Properties of the Turkish Version of Young Children's Participation and Environment Measure (YC-PEM) in Young Children With Typical Development and Neurodevelopmental Disorders
Brief Title: Psychometric Properties of the Turkish Version of Young Children's Participation and Environment Measure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Seyhan, Dr.Pt, Hacettepe University
Other Study IDs: GO 21/430 2021/07-44
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Child Development Disorder; Activity, Motor
Keywords: Cerebral palsy; Activity; Participaiton; Environment
MeSH Terms: conditions — Developmental Disabilities; Motor Activity; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Children under five years old

SUMMARY:
The Young Children's Participation and Environment Measure (YC-PEM) is a parent/caregiver reported outcome measure that evaluates the participation status and environmental factors of children under five years old. The aim of this study is to translate the Young Children's Participation and Environment Measure (YC-PEM) into the Turkish language and to investigate the psychometric properties of the Turkish version of YC-PEM in children with typical development and neurodevelopmental disabilities under five years old.

DETAILED DESCRIPTION:
Cross-cultural adaptation Rest-retest reliability Discriminant validity Concurrent validity

ELIGIBILITY:
Inclusion Criteria:

* children under five years
* children with neurodevelopmental disabilities

Exclusion Criteria:

* parents who refused to participate in the study

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with typical development and children with neurodevelopmental disabilities (Cerebral palsy, obstetric brachial plexus palsy, autism spectrum disorders or developmental coordination disorders etc.)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Young children's participation and environment measure (YC- PEM) | two years
  Young children's participation and environment measure (YC- PEM) is developed for assessing the activity and participation levels and effects of environmental factors on functional abilities in children with neurodevelopmental disabilities or typically development under five years.

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | two years
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing the activity and participation levels and effects of environmental factors on functional abilities in children with neurodevelopmental disabilities or typically development under seven years.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra S Bıyık, Principal Investigator — Dr.Pt
Locations (1):
- Hacettepe University, Ankara, Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided